CLINICAL TRIAL: NCT02739620
Title: Alternative Exercise Program to Improve Skeletal Muscle Function and Fatigue in Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Michael J. Toth, Ph.D., Associate Professor of Medicine, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: M16-333
Record Dates: First submitted 2016-04-08; First posted 2016-04-15 (Estimated); Results first posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- NMES (Experimental): Neuromuscular electrical stimulation (NMES) group
  Interventions: Device: Neuromuscular electrical stimulation
- Control (No Intervention): Control group

INTERVENTIONS:
Device: Neuromuscular electrical stimulation — Neuromuscular electrical stimulation will be performed 5 times/week for one hour each day for 2 months.
  Arms: NMES

SUMMARY:
Exercise training has beneficial effects in cancer survivors to minimize some of the side effects of cancer and its treatment and improve long-term prognosis, but there are numerous hurdles for individuals diagnosed with, and being treated for, cancer to participate in exercise programs. The goal of this research study is to begin to evaluate whether exercise training via neuromuscular electrical stimulation (NMES) has beneficial effects on skeletal muscle size and function in cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

1. stage I, II or III breast cancer
2. receiving neoadjuvant or adjuvant chemotherapy with or without radiation
3. a body mass index <35 kg/m2.

Exclusion Criteria:

1. metastatic disease, a prior history of cancer, excluding non-melanoma skin cancer, or prior receipt of chemotherapy
2. autoimmune, vascular or neuromuscular disease that could alter skeletal muscle
3. prior knee or hip replacement
4. contraindications for use of neuromuscular electrical stimulation, including an implanted cardiac defibrillator or pacemaker, lower extremity blood clot or coagulopathy
5. pregnancy

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2019-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Toth, PhD, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont College of Medicine, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: Yes
Research data (deidentified) which documents, supports and validates research findings will be stored on the University of Vermont College of Medicine computer system and will be made available upon final acceptance for publication of the major findings from the proposed studies. This includes raw data generated from all clinical and laboratory-based assessments under a data-sharing agreement.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NMES | Control
Started | 12 | 10
Baseline Testing | 12 | 10
Intervention Phase | 10 | 10
Post-intervention Testing | 9 | 8
Completed | 9 | 8
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 3 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NMES | Control | Total
Number analyzed (Participants) | 12 | 10 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (5.5) | 55.5 (8.8) | 54.5 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 11 | 9 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 10 | 22
Weight [Mean (Standard Deviation); unit: kilograms] | 75.0 (15.1) | 71.2 (14.2) | 73.2 (14.5)
Height [Mean (Standard Deviation); unit: centimeters] | 163.4 (10.5) | 161.6 (6.9) | 162.6 (8.8)
Percentage of body fat [Mean (Standard Deviation); unit: percent] | 42.4 (7) | 39.9 (5.9) | 41.3 (6.5)
Fat mass [Mean (Standard Deviation); unit: kilograms] | 31.9 (10.6) | 28.3 (8.8) | 30.2 (9.8)
Fat-free mass [Mean (Standard Deviation); unit: kilograms] | 41.5 (5.4) | 41.3 (6.4) | 41.4 (5.7)
Appendicular skeletal muscle mass [Mean (Standard Deviation); unit: kilograms] | 25.3 (3.9) | 24.7 (5.2) | 25.0 (4.4)

OUTCOME MEASURES:

1. Primary Outcome: Maximal Calcium-activated Tension Single Muscle Fiber Tension
Description: Tension (force per unit muscle fiber cross-sectional area) from segments of chemically-skinned single human muscle fibers will be assessed under maximal calcium-activated condition, with muscle fiber type determined post-measurement by gel electrophoresis
Time Frame: Difference between values at baseline at 2 months
Population: The sample sizes reflect the number of volunteers with paired data at both baseline and 2-month testing.
Measure: Mean (Standard Error); unit: milliNewtons per millimeter^2
Arm/Group | NMES | Control
Number analyzed (Participants) | 9 | 8
milliNewtons per millimeter^2
  Baseline testing | 185 (10) | 172 (10)
  Post-intervention testing | 172 (9) | 168 (10)

2. Primary Outcome: Cross-sectional Area of Skeletal Muscle Fibers
Description: Cross-sectional area of skeletal muscle fibers will be evaluated using immunohistochemistry, with specification of all relevant muscle fiber types
Time Frame: Difference between values at baseline at 2 months
Population: The sample sizes reflect the number of volunteers with paired data at both baseline and 2-month testing.
Measure: Mean (Standard Error); unit: micrometers^2
Arm/Group | NMES | Control
Number analyzed (Participants) | 9 | 8
micrometers^2
  Baseline testing | 2432 (246) | 2320 (261)
  Post-intervention testing | 2694 (246) | 2381 (260)

3. Primary Outcome: Intermyofibrillar Mitochondrial Content
Description: Area fraction of intermyofibrillar mitochondria will be assessed by electron microscopy
Time Frame: Difference between values at baseline at 2 months
Population: The sample sizes reflect the number of volunteers with paired data at both baseline and 2-month testing and the fact that electron microscopy measures could not be completed on one volunteer because of insufficient muscle tissue.
Measure: Mean (Standard Error); unit: percentage of image area
Arm/Group | NMES | Control
Number analyzed (Participants) | 9 | 7
percentage of image area
  Baseline testing | 2.72 (0.24) | 2.62 (0.26)
  Post-intervention testing | 2.75 (0.25) | 2.56 (0.26)

4. Secondary Outcome: Single Muscle Fiber Contractile Velocity
Description: Single muscle fiber contractile velocity assessed using isotonic load clamps, with muscle fiber type determined post-measurement by gel electrophoresis. The velocity of contraction is expressed relative to the length of the muscle fiber segment evaluated (as measured using a eyepiece micrometer during assessments) per second.
Time Frame: Difference between values at baseline at 2 months
Population: The sample sizes reflect the number of volunteers with paired data at both baseline and 2-month testing.
Measure: Mean (Standard Error); unit: muscle lengths per second
Arm/Group | NMES | Control
Number analyzed (Participants) | 9 | 8
muscle lengths per second
  Baseline testing | 2.1 (0.08) | 1.92 (0.09)
  Post-intervention testing | 1.92 (0.9) | 1.73 (0.8)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | NMES | Control
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/10
Other Adverse Events (participants affected / at risk) | 0/12 | 1/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NMES (N=12) | Control (N=10)
Hospitalization (Infections and infestations) | 0 (0) | 1 (1) — Hospitalization for pyelonephritis. Adjudicated to be severe, unexpected and not related to study participation.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NMES (N=12) | Control (N=10)
Febrile episode (Infections and infestations) | 0 (0) | 1 (1) — Patient became febrile during testing. Adjudicated to be moderate severity, unexpected and not related to study participation/intevention.

LIMITATIONS AND CAVEATS:
Our study was powered to detect effects on skeletal muscle at the cellular level over a short time period during treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-15): https://cdn.clinicaltrials.gov/large-docs/20/NCT02739620/Prot_SAP_000.pdf